CLINICAL TRIAL: NCT05133570
Title: Study Evaluating the Effectiveness of Treatment With Vista Care®, in Arterial Ulcers of the Lower Extremities
Acronym: VISTA CARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0312
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Wound Heal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: vista care — Prospective, open-label, multi-centre study evaluating the performance of the VistaCare® wound healing device in routine practice.

SUMMARY:
The prevalence of chronic wounds is around 2 million people in France per year. A chronic wound is a wound that has been evolving for more than 6 weeks. The main causes are: venous causes, arterial causes and microcirculatory causes. In some aetiologies (particularly arterial causes), there is no radical therapeutic solution (no possibility of revascularisation) and the wounds are often difficult to treat and may even eventually lead to amputation. The recommendations for treating wounds are (in addition to carrying out an etiological treatment when possible) to carry out mechanical detersion and to maintain a moist wound environment. In addition to various medical devices such as dressings, adjuvant treatments that are not specific to the etiology of the wound, such as electrotherapy, negative pressure therapy or other devices such as the VistaCare®, are indicated in France.

DETAILED DESCRIPTION:
Prospective, open-label, multi-centre study evaluating the performance of the VistaCare® wound healing device in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* -Patient able and willing to comply with the requirements of the including hospitalization for up to 15 days.
* Patient whose wound to be studied is located in a location compatible with the use of VistaCare®, namely the leg including the knee but excluding the upper thigh
* Agreement of the study no-objection form
* Age greater than or equal to 18 years
* Patient affiliated to a social security scheme

Exclusion Criteria:

* -Patient with general signs of infection at the time of inclusion (fever, lymphangitis, pus ...). Patient with active smoking Subject under guardianship or deprived of liberty Failure to obtain patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient whose wound to be studied is located in a location compatible with the use of VistaCare®, namely the leg including the knee but excluding the upper thigh with arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2023-10-29 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the healing performance of the VistaCare® device in routine practice in patients with chronic arterial leg wounds. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- BLAISE, Grenoble, France